CLINICAL TRIAL: NCT07023328
Title: BalL Exercises tO Prevent FrAilty in OldeR ADults (LEOPARD): A Pragmatic, Open-label, Randomized Controlled Trial.
Brief Title: BalL Exercises tO Prevent FrAilty in OldeR ADults (LEOPARD)
Acronym: (LEOPARD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIO-2023-0255
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ball Exercise Group (Experimental): Participants in this arm are pre-frail older adults who will undergo a structured ball exercise program
  Interventions: Behavioral: A structured ball exercise program
- Usual Care Group (No Intervention): Participants in this arm are pre-frail older adults who will usual care

INTERVENTIONS:
Behavioral: A structured ball exercise program — Pre-frail older adults will undergo a structured ball exercise program
  Arms: Ball Exercise Group

SUMMARY:
This study aims to examine the effects of a multi-component intervention incorporating Swiss ball exercises and nutritional counseling on reducing frailty in a sample of pre-frail older adults in primary care. It also aims to assess its effects on physical performance, functional status, and cognitive and well-being measures.

Participants aged between 65 and 75 years will be randomly assigned to the intervention group and "usual care" group .

Over a 3-month period, the multi-component intervention will consist of Swiss ball exercises and nutritional counseling, whereas the "usual care" group will get verbal general health counseling on healthy eating and physical activity recommendations.

Outcome Assessors who are blinded to treatment allocation will evaluate primary and secondary outcomes at the end of the intervention (3 months), and after 6 months follow-up period.

ELIGIBILITY:
Inclusion Criteria

* Age between 65 and 75 years
* Pre-frail status according to the FRAIL Scale assessment
* Ability to rise from a chair without assistance
* Ability to perform the Apley scratch test
* Ability to bend forward without significant pain

Exclusion Criteria

* Hospitalization within the past 3 months
* Currently receiving oxygen therapy
* Congestive heart failure (CHF) with an ejection fraction less than 25%
* Severe aortic stenosis
* Uncontrolled paroxysmal vertigo
* Active neoplastic disease or terminal illness
* Severe cognitive impairment
* Neurological disorders (e.g., Parkinson's disease, multiple sclerosis)
* Bedridden status
* Major disability or mobility disorder
* Chest pain at rest, during activities, or with physical exertion
* History of loss of consciousness within the past 12 months
* Medical advice to avoid vigorous physical activity

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
FRAIL scale | Measurements will be assessed at baseline (before randomization) after 3 months at the end of the intervention, and after 6 months follow-up period.
  The FRAIL scale will be used to measure the participants' frailty status as the primary outcome.
  The FRAIL scale is an interview-based 5-item instrument that measures the level of frailty. It does not need physical performance measures. The items measure components of fatigue (self report), resistance (difficulty walking up 10 steps without resting), ambulation (difficulty walking 300 m), unintentional weight loss (>5% in the past year), and illnesses (≥5 chronic conditions).
  The FRAIL scale scores range from 0-5 ((i.e., 1 point for each component; 0=best to 5=worst) and represents frail (3-5), prefrail (1-2), and robust (0) health states .

SECONDARY OUTCOMES:
Grip strength measurement | Measurements will be assessed at baseline (before randomization) after 3 months at the end of the intervention, and after 6 months follow-up period.
  Physical performance measures will be conducted. Upper muscle strength will be measured using the grip strength measurement. Maximum grip strength of the dominant hand (in kg) will be measured during vital signs measurements using a Jamar digital dynamometer grip. Grip strength in kilograms will be measured using a standardized protocol; participants will be seated with the ipsilateral shoulder adducted and neutrally rotated, the elbow flexed to 90 degrees, and the forearm and wrist neutrally positioned. The participants will be asked to perform three maximum force trials with their dominant hand interspersed by 1 minute and the highest measure observed will be observed.
The Five Times Sit to Stand Test (5TSTS) | Measurements will be assessed at baseline (before randomization) after 3 months at the end of the intervention, and after 6 months follow-up period.
  Physical performance measures will be conducted. Lower limb strength will be measured using the Five Times Sit to Stand Test (5TSTS).Participants will be instructed to rise as quickly as possible from a seated position, with full body weight on the chair, to a standing posture, with their legs fully extended, while keeping their arms folded across their chest. The 5TSTS measures the time taken, in seconds, to complete five repeated chair stands. The test performance will be based on its duration; consequently, the shorter time taken by the patient, the better their functional condition would be.
The 4-m gait speed (4MGS) | Measurements will be assessed at baseline (before randomization) after 3 months at the end of the intervention, and after 6 months follow-up period.
  To perform the test, a flat unobstructed course will be identified and 4 m marked out with tape. The participant will be positioned with the toes just touching the start line. The following standardized instructions will be given: "This is our walking course. I want you to walk to the other end of the course at your usual speed, just as if you were walking down the street to go to the shops. Walk all the way past the other end of the tape before you stop. Ready…begin". Timing with a stopwatch will be started when the participant begins to move, not on the command "begin". Timing will be stopped when the participant's first foot completely crosses the 4-m line. The walk test will be repeated without rest and the faster of the two times will be used to calculate the 4MGS, expressed in m·s-1. Participants will be allowed to use their normal walking aids (e.g. cane).
The Timed Up and Go test (TUG) | Measurements will be assessed at baseline (before randomization) after 3 months at the end of the intervention, and after 6 months follow-up period.
  The participant will be asked to sit on a chair (chair height=45cm) with an upright posture, feet placed flat on the ground, and arms crossed on their chest. Next, participants will be instructed to rise from the chair, walk to, and around a cone (three meters) in front of them, walk back to the chair, and return to the starting position. Time will be recorded starting the moment the participant's back loses contact with the chair and concluded when the starting position is regained. A score of ≥ 14 seconds has been shown to indicate reduced mobility, impaired balance, and a high risk of falls.
Lawton's Instrumental Activities of Daily Living (IADL) Scale | Measurements will be assessed at baseline (before randomization) after 3 months at the end of the intervention, and after 6 months follow-up period.
  Functional status will be assess using the Lawton's Instrumental Activities of Daily Living (IADL) Scale). The Lawton IADL Scale takes approximately 10 to 15 minutes to administer. It contains 8 items that are rated with a summary score from 0 (low functioning) to 8 (high functioning). For men, the areas of food preparation, housekeeping, and laundering will be excluded. Participants are scored according to their highest level of functioning in that category. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 to 5 for men.
The Montreal Cognitive Assessment (MoCA) | Measurements will be assessed at baseline (before randomization) after 3 months at the end of the intervention, and after 6 months follow-up period.
  Cognitive function will be measured using the Montreal Cognitive Assessment (MoCA). The MoCA test is conducted over 20 minutes to measure seven cognitive domains, including executive functions, naming, verbal memory registration and learning, attention, abstraction, delay recall memory, and orientation. MoCA scores range from 0 to 30, higher scores reflect good global cognitive function.
Patient Health Questionnaire-4' (PHQ-4) | Measurements will be assessed at baseline (before randomization) after 3 months at the end of the intervention, and after 6 months follow-up period.
  PHQ-4 will be used to screen for depression and anxiety. PHQ-4 is a 4-item inventory rated on a 4-point Likert-type scale with response options including the following: not at all (score = 0), several days (score = 1), more than half the days (score = 2), and nearly every day (score = 3). PHQ-4 scores will be computed by adding scores on individual items. PHQ-4 scores determine 'Severe' (score range 9-12), 'Moderate' (6-8), 'Mild' (3-5), and 'Normal' (0-2) risk of anxiety or depression. On each subscale, a score of 3 or greater is considered a risk for anxiety or depression.
World Health Organization Well-Being Index (WHO-5) | Measurements will be assessed at baseline (before randomization) after 3 months at the end of the intervention, and after 6 months follow-up period.
  The 5-item World Health Organization Well-Being Index (WHO-5) is a short questionnaire covering five positively worded items, related to positive mood (good spirits, relaxation), vitality (being active and waking up fresh and rested), and general interests (being interested in things). Each of the five items in the WHO-Five is rated on a 6-point Likert scale from 0 (not present) to 5 (constantly present). The raw score ranges from 0 to 25, and the percentage final score (0-100%) can be obtained by multiplying the result by 4. A cutoff of <13 (or <50%) indicates poor psychological well-being.